CLINICAL TRIAL: NCT03271060
Title: Comparative Study Between Posterior Lumbar Interbody Fusion(PLF) and Intertransverse Process Fusion in Treatment of Spodylolithesis
Brief Title: Comparative Study Between Posterior Lumbar Interbody Fusion(PLIF) and Intertransverse Process Fusion in Treatment of Spodylolithesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Garamoun Abd El Zaher, Doctor, Assiut University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lumbar spondylolisthesis
Record Dates: First submitted 2017-08-31; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Lumbar Spondylolisthesis
MeSH Terms: conditions — Spondylolisthesis

STUDY DESIGN:
Intervention Model Description: Posterior inter body fusion and inter transverse process bone graft
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbar spondylolisthesis1 (Active Comparator)
  Interventions: Procedure: Inter transverse bone grafting
- Lumbar spondylolisthesis 2 (Active Comparator)
  Interventions: Procedure: Posterior lumbar interbody fusion

INTERVENTIONS:
Procedure: Posterior lumbar interbody fusion — Lumbar fusion by screws and inter vertebral cage
  Arms: Lumbar spondylolisthesis 2
Procedure: Inter transverse bone grafting — Inter transverse process bone grafting by bone graft from illiac crest or other sites
  Arms: Lumbar spondylolisthesis1

SUMMARY:
The first technique described for interbody fusion was the anterior lumbar interbody fusion (ALIF).(20) For this technique, the intervertebral disc is accessed through a retroperitoneal or transperitoneal approach.

While the posterior approach was first described by Russell Hibbs in 1911, in the 1950's, Cloward (7)popularized the posterior approach for a posterior lumbar interbody fusion (PLIF).

DETAILED DESCRIPTION:
In this study we will try to identify the benefits and outcome of posterior lumbar interbody fusion and inter transverse process bone graft fusion.

ELIGIBILITY:
Inclusion Criteria:

* lumbar spondylolisthesis

Exclusion Criteria:

* infection of lumbar spine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-08-30 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Back pain | 1year postoperative
  Back pain severity grading mild, moderate, severe